CLINICAL TRIAL: NCT04271358
Title: Peer Coaching Adaptive Self-Management Interventions for Young Adults With Congenital Heart Disease
Brief Title: Peer Coaching Intervention in Young Adults With Congenital Heart Disease
Acronym: CHASM in ACHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Adult Congenital Heart Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00103600
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Congenital Heart Disease; Congenital Heart Defect
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Once enrolled, participants will be randomly assigned to the intervention or control group (1:1 ratio)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Coaching (Experimental): Participant receive a 6 month peer health coaching intervention.
  Interventions: Behavioral: Peer Health Coaching
- Education only (No Intervention): Participants receive education-only material (newsletter) biweekly for 6 months

INTERVENTIONS:
Behavioral: Peer Health Coaching — The Peer Coaching group will receive 6 months of peer health coaching via a secure telephone and text messaging system.
  Arms: Peer Coaching

SUMMARY:
The purpose of the study is to evaluate a peer coaching intervention in young adults with congenital heart disease.

DETAILED DESCRIPTION:
Our research team has developed a peer coaching intervention that has been deployed to promote activated self-management for AYAs with several conditions, and this has been modified adolescents and young adults (AYA) with with congenital heart disease (CHD). This study will be conducted over two years and pair AYA with CHD with a peer coach who also has CHD has successfully navigated the transition to adult medical care and over six months will work to promote the motivation for self-care as well as the development of self-management skills. This pilot study will test feasibility and acceptability, as well as preliminary efficacy and long-term effects on successful transfer to adult cardiology.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-26
* Diagnosis of congenital heart disease
* Patient at a Duke pediatric cardiology clinic
* Access to a smart phone

Exclusion Criteria:

* Cognitive delay
* Patient at an adult cardiology clinic

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2032-03-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate number of participants enrolled | Up to 2 months after recruitment closes
  Evaluate the number of participants contacted about the study who actually enrolled
Evaluate completion of study | Up to 8 months after enrollment of each participant
  Determine the number of participants who enrolled in the study who completed it
Measure impact on health | Up to 8 months after enrollment of each participant
  Evaluate the number of participant who stated the intervention had a positive impact on their health
Determine change in patient activation | baseline, 3 months, 6 months
  Determine change in patient activation as measured by changes over time on the Patient Activation Measure (PAM)
Determine change in self-management | baseline, 3 months, 6 months
  Determine change in self-management as measured by changes over time in the Partners in health Scale (PIH)

SECONDARY OUTCOMES:
Determine change in transition readiness | baseline, 3 months, 6 months
  Determine the change in transition readiness over 6 months as measured by the Transition Readiness Assessment Questionaire (TRAQ)
Determine change in health related quality of life | baseline, 3 months, 6 months
  Determine the change in health related quality of life over 6 months as measured by the Short-From 12 (SF-12)
Determine change in emotional health | baseline, 3 months, 6 months
  Determine the change in emotional health over 6 months as measured by the Brief Symptom Inventory (BSI)
Evaluate successful transfer of participants from pediatric to adult cardiology care | up to 10 years
  Evaluate number of participants that transfer from pediatric to adult cardiology care with at least consecutive visits 10 years post study

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Krasuski, MD, Principal Investigator — Duke University; Gary Maslow, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke Health, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No